CLINICAL TRIAL: NCT02780024
Title: Metformin and Neo-adjuvant Temozolomide and Hypofractionated Accelerated Limited-margin Radiotherapy Followed by Adjuvant Temozolomide in Patients With Glioblastoma Multiforme (M-HARTT STUDY)
Brief Title: Metformin, Neo-adjuvant Temozolomide and Hypo- Accelerated Radiotherapy Followed by Adjuvant TMZ in Patients With GBM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, George Shenouda, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUHC ID: 4315
Record Dates: First submitted 2015-05-20; First posted 2016-05-23 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma Multiforme
Keywords: Neo-Adjuvant Metformin; Neo-Adjuvant Temozolomide; Temozolomide and accelerated hypofractionation; Metformin and accelerated hypofractionation; Adjuvant Temozolomide; Adjuvant Metformin
MeSH Terms: conditions — Glioblastoma | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Registered one arm study (Experimental): Two weeks of neo-adjuvant Metformin+Temozolomide followed by accelerated hypofractionation using an IMRT technique+TMZ & Metformin followed by TMZ, and Metformin as adjuvant component.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin,
  Other Names: Glucophage

SUMMARY:
Glioblastoma Multiforme is one of the most common, and unfortunately one of the most aggressive brain tumors in adults with most of the patients recurring and dying of the disease with a median survival of 16 months from diagnosis.

Current treatment for patients with newly diagnosed Glioblastoma Multiforme (GBM) is safe maximal surgical resection followed by concomitant conventional Radiotherapy (RT) delivered in 6 weeks + Temozolomide (TMZ) followed by TMZ for 6 to 12 cycles.

Recent scientific research has shown that Metformin, a common drug used to treat diabetes mellitus, may improve the results of the treatment in patients with a variety of cancers, such as breast, colon, and prostate cancer. Metformin is an attractive and safe medication to be used in this group of patients because of its very low toxicity.

In our center the investigators have been using TMZ for 2 weeks prior to a short course (4 weeks) of RT which equivalent to the standard RT of 6 weeks. Temozolomide is used 2 weeks before RT + TMZ, and this is followed by the 6 to 12 cycles of TMZ. Our results are quiet encouraging with a median survival of 20 months, and acceptable toxicity.

DETAILED DESCRIPTION:
Metformin, a drug with a very safe toxicity profile, is an attractive molecule to be tested in patients with newly diagnosed GBM in a phase I clinical trial. This is based on its potential to inhibit the proliferation of GBM CSCs through its mechanism of action which is similar to IR and TMZ. Metformin, IR, and TMZ stimulate AMPK leading to the subsequent inhibition of cellular proliferation. Therefore, it is hypothesized that the addition of Metformin to concomitant IR and TMZ may increase the efficiency of IR and TMZ, which are currently considered as the standard of care for patients with GBM. In addition, Metformin lowers blood glucose levels, and subsequently reduces the insulin and Insulin-Growth-factors which are growth-promoting factors with a direct impact on GBM cellular proliferation and invasion.

Metformin may improve the outcomes of patients with GBM when added to current treatment consisting of maximal safe surgical resection followed by neo-adjuvant TMZ and concomitant accelerated hypofractionated limited-margin XRT followed by adjuvant TMZ. Our Neuro-Oncology group at McGill University reviewed the results of an ongoing Phase II study in patients with GBM. A group of 33 patients were treated according to protocol, and with a median follow-up of 11 months, the median survival was 17.5 months which compares favourably to current results from standard treatment with a beneficial 2-week shortening of the XRT treatment time.

This is a phase II clinical trial to assess the feasibility and overall toxicity of adding Metformin to Neoadjuvant Temozolomide followed by concomitant Temozolomide and accelerated hypofractionated limited-margin radiotherapy and followed by adjuvant Temozolomide in patients with newly diagnosed GBM.

It is expected that the proposed study treatment will improve the median survival from current values of 20 months (current MUHC Neo-adjuvant Phase 2 data) to 25 months. This means an improved outcome of 25%. Using one-tailed statistics, and with a power of 0.8 and an alpha of 0.05, the sample size for this Phase II trial will be 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Histological confirmation of supra-tentorial GBM
* KPS > 60
* Neurological function 0 or 1
* Adequate bone marrow as defined below:

Absolute neutrophil count (ANC) ≥ 1500 cells/mm3. Platelets ≥ 100,000 cells/mm3 Hemoglobin ≥ 10 g/dl.

* Adequate renal function, as defined below:
* Creatinine clearance of >60 ml/min/1.73m2 (using the Cockcroft Gault equation for eGFR) within 14 days prior to study registration
* Adequate hepatic function, as defined below:
* Bilirubin of 1.7 to 18.9 umol/L within 14 days prior to study registration
* ALT ≤ 3 x normal range within 14 days prior to study registration
* Neo-adjuvant TMZ and Metformin to start within 4 weeks of surgery
* Concomitant TMZ and Metformin and accelerated Hypofractionated EBRT to start at least 2 weeks after adjuvant TMZ starting date, and no later than five weeks from surgery.
* Surgical diagnosis/intervention may include: partial or near total resection
* Patients must have recovered from the effects of surgery, postoperative infection and other complications before study registration.
* A diagnostic contrast-enhanced MRI or CT scan of the brain must be performed preoperatively and postoperatively. The postoperative scan must be done within 28 days prior to the initiation of neo-adjuvant TMZ. Preoperative and postoperative scans must be the same type. Patients unable to undergo MR imaging can be enrolled provided pre- and post-operative contrast-enhanced CT scans are obtained and are of sufficient quality.
* History/physical examination, including neurologic exam within 14 days prior to study registration.
* Documentation of steroid doses within 14 days prior to study registration and stable or decreasing steroid dose within 5 days prior to registration.
* For females of child-bearing potential, negative serum pregnancy test within 72hours prior to starting TMZ and Metformin. Women of childbearing potential and male participants must practice adequate contraception.
* Adequate tissue specimen for MGMT status analysis.
* Able to sign an informed study-specific consent

Exclusion Criteria:

* Diabetic patients both type I and type II.
* No tissue provided for MGMT promoter methylation status determination.
* Margin of contrast-enhanced residual mass closer than 15 mm from the optic chiasm or optic nerves.
* Prior invasive malignancy (except for non-melanoma skin cancer) unless disease free for ≥ 3 years
* Recurrent or multifocal GBM.
* Prior chemotherapy or radio-sensitizers for cancers of the head and neck region; prior chemotherapy for a different cancer is allowable.
* Severe, active co-morbidity, defined as follows:

  * Acute or chronic renal failure.
  * Unstable angina and/or congestive heart failure requiring hospitalization
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition.
  * Major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
  * Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
  * Pregnant or lactating women, due to possible adverse effects on the developing foetus or infant due to study drug.
  * Prior allergic reaction to Temozolomide or Metformin.
  * Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2021-10-20 (Actual); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients completing the study treatment | At one year
  To determine overall survival

SECONDARY OUTCOMES:
To assess toxicity of the regimen | One year
  Toxicity will be assessed and graded according to CTCAE-V4

CONTACTS AND LOCATIONS:
Overall Officials: George Shenouda, M.D., Principal Investigator — Radiation Oncologist
Locations (1):
- Montreal Neurological Institute - McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Alcantara Llaguno SR, Chen Y, McKay RM, Parada LF. Stem cells in brain tumor development. Curr Top Dev Biol. 2011;94:15-44. doi: 10.1016/B978-0-12-380916-2.00002-4. PMID 21295683
- [Background] Singh SK, Clarke ID, Terasaki M, Bonn VE, Hawkins C, Squire J, Dirks PB. Identification of a cancer stem cell in human brain tumors. Cancer Res. 2003 Sep 15;63(18):5821-8. PMID 14522905
- [Background] Singh SK, Hawkins C, Clarke ID, Squire JA, Bayani J, Hide T, Henkelman RM, Cusimano MD, Dirks PB. Identification of human brain tumour initiating cells. Nature. 2004 Nov 18;432(7015):396-401. doi: 10.1038/nature03128. PMID 15549107
- [Background] He J, Shan Z, Li L, Liu F, Liu Z, Song M, Zhu H. Expression of glioma stem cell marker CD133 and O6-methylguanine-DNA methyltransferase is associated with resistance to radiotherapy in gliomas. Oncol Rep. 2011 Nov;26(5):1305-13. doi: 10.3892/or.2011.1393. Epub 2011 Jul 18. PMID 21769436
- [Background] Metellus P, Nanni-Metellus I, Delfino C, Colin C, Tchogandjian A, Coulibaly B, Fina F, Loundou A, Barrie M, Chinot O, Ouafik L, Figarella-Branger D. Prognostic impact of CD133 mRNA expression in 48 glioblastoma patients treated with concomitant radiochemotherapy: a prospective patient cohort at a single institution. Ann Surg Oncol. 2011 Oct;18(10):2937-45. doi: 10.1245/s10434-011-1703-6. Epub 2011 Apr 9. PMID 21479688
- [Background] Ben Sahra I, Le Marchand-Brustel Y, Tanti JF, Bost F. Metformin in cancer therapy: a new perspective for an old antidiabetic drug? Mol Cancer Ther. 2010 May;9(5):1092-9. doi: 10.1158/1535-7163.MCT-09-1186. Epub 2010 May 4. PMID 20442309
- [Background] Evans JM, Donnelly LA, Emslie-Smith AM, Alessi DR, Morris AD. Metformin and reduced risk of cancer in diabetic patients. BMJ. 2005 Jun 4;330(7503):1304-5. doi: 10.1136/bmj.38415.708634.F7. Epub 2005 Apr 22. No abstract available. PMID 15849206
- [Background] Murtola TJ, Tammela TL, Lahtela J, Auvinen A. Antidiabetic medication and prostate cancer risk: a population-based case-control study. Am J Epidemiol. 2008 Oct 15;168(8):925-31. doi: 10.1093/aje/kwn190. Epub 2008 Aug 11. PMID 18700234
- [Background] Bolster DR, Crozier SJ, Kimball SR, Jefferson LS. AMP-activated protein kinase suppresses protein synthesis in rat skeletal muscle through down-regulated mammalian target of rapamycin (mTOR) signaling. J Biol Chem. 2002 Jul 5;277(27):23977-80. doi: 10.1074/jbc.C200171200. Epub 2002 May 7. PMID 11997383
- [Background] Ben Sahra I, Laurent K, Loubat A, Giorgetti-Peraldi S, Colosetti P, Auberger P, Tanti JF, Le Marchand-Brustel Y, Bost F. The antidiabetic drug metformin exerts an antitumoral effect in vitro and in vivo through a decrease of cyclin D1 level. Oncogene. 2008 Jun 5;27(25):3576-86. doi: 10.1038/sj.onc.1211024. Epub 2008 Jan 21. PMID 18212742
- [Background] Zhuang Y, Miskimins WK. Cell cycle arrest in Metformin treated breast cancer cells involves activation of AMPK, downregulation of cyclin D1, and requires p27Kip1 or p21Cip1. J Mol Signal. 2008 Dec 1;3:18. doi: 10.1186/1750-2187-3-18. PMID 19046439
- [Background] Wang LW, Li ZS, Zou DW, Jin ZD, Gao J, Xu GM. Metformin induces apoptosis of pancreatic cancer cells. World J Gastroenterol. 2008 Dec 21;14(47):7192-8. doi: 10.3748/wjg.14.7192. PMID 19084933
- [Background] Hirsch HA, Iliopoulos D, Tsichlis PN, Struhl K. Metformin selectively targets cancer stem cells, and acts together with chemotherapy to block tumor growth and prolong remission. Cancer Res. 2009 Oct 1;69(19):7507-11. doi: 10.1158/0008-5472.CAN-09-2994. Epub 2009 Sep 14. PMID 19752085
- [Background] Jiralerspong S, Palla SL, Giordano SH, Meric-Bernstam F, Liedtke C, Barnett CM, Hsu L, Hung MC, Hortobagyi GN, Gonzalez-Angulo AM. Metformin and pathologic complete responses to neoadjuvant chemotherapy in diabetic patients with breast cancer. J Clin Oncol. 2009 Jul 10;27(20):3297-302. doi: 10.1200/JCO.2009.19.6410. Epub 2009 Jun 1. PMID 19487376
- [Background] Micic D, Cvijovic G, Trajkovic V, Duntas LH, Polovina S. Metformin: its emerging role in oncology. Hormones (Athens). 2011 Jan-Mar;10(1):5-15. doi: 10.14310/horm.2002.1288. PMID 21349801
- [Background] Libby G, Donnelly LA, Donnan PT, Alessi DR, Morris AD, Evans JM. New users of metformin are at low risk of incident cancer: a cohort study among people with type 2 diabetes. Diabetes Care. 2009 Sep;32(9):1620-5. doi: 10.2337/dc08-2175. Epub 2009 Jun 29. PMID 19564453
- [Background] Kumar S, Meuter A, Thapa P, Langstraat C, Giri S, Chien J, Rattan R, Cliby W, Shridhar V. Metformin intake is associated with better survival in ovarian cancer: a case-control study. Cancer. 2013 Feb 1;119(3):555-62. doi: 10.1002/cncr.27706. Epub 2012 Dec 3. PMID 23208739
- [Background] Zhang WB, Wang Z, Shu F, Jin YH, Liu HY, Wang QJ, Yang Y. Activation of AMP-activated protein kinase by temozolomide contributes to apoptosis in glioblastoma cells via p53 activation and mTORC1 inhibition. J Biol Chem. 2010 Dec 24;285(52):40461-71. doi: 10.1074/jbc.M110.164046. Epub 2010 Sep 29. PMID 20880848
- [Background] Wurth R, Pattarozzi A, Gatti M, Bajetto A, Corsaro A, Parodi A, Sirito R, Massollo M, Marini C, Zona G, Fenoglio D, Sambuceti G, Filaci G, Daga A, Barbieri F, Florio T. Metformin selectively affects human glioblastoma tumor-initiating cell viability: A role for metformin-induced inhibition of Akt. Cell Cycle. 2013 Jan 1;12(1):145-56. doi: 10.4161/cc.23050. Epub 2012 Dec 19. PMID 23255107
- [Background] Sato A, Sunayama J, Okada M, Watanabe E, Seino S, Shibuya K, Suzuki K, Narita Y, Shibui S, Kayama T, Kitanaka C. Glioma-initiating cell elimination by metformin activation of FOXO3 via AMPK. Stem Cells Transl Med. 2012 Nov;1(11):811-24. doi: 10.5966/sctm.2012-0058. Epub 2012 Nov 15. PMID 23197693
- [Background] Ferla R, Haspinger E, Surmacz E. Metformin inhibits leptin-induced growth and migration of glioblastoma cells. Oncol Lett. 2012 Nov;4(5):1077-1081. doi: 10.3892/ol.2012.843. Epub 2012 Aug 3. PMID 23162655
- [Background] Bao S, Wu Q, McLendon RE, Hao Y, Shi Q, Hjelmeland AB, Dewhirst MW, Bigner DD, Rich JN. Glioma stem cells promote radioresistance by preferential activation of the DNA damage response. Nature. 2006 Dec 7;444(7120):756-60. doi: 10.1038/nature05236. Epub 2006 Oct 18. PMID 17051156
- [Background] Bleau AM, Holland EC. [Chemotherapeutic treatment of gliomas increases the amount of cancer stem-like cells]. Med Sci (Paris). 2009 Oct;25(10):775-7. doi: 10.1051/medsci/20092510775. No abstract available. French. PMID 19849969
- [Background] Lu H, Li Y, Shu M, Tang J, Huang Y, Zhou Y, Liang Y, Yan G. Hypoxia-inducible factor-1alpha blocks differentiation of malignant gliomas. FEBS J. 2009 Dec;276(24):7291-304. doi: 10.1111/j.1742-4658.2009.07441.x. PMID 19912340
- [Background] Al-Hajj M, Clarke MF. Self-renewal and solid tumor stem cells. Oncogene. 2004 Sep 20;23(43):7274-82. doi: 10.1038/sj.onc.1207947. PMID 15378087
- [Background] Dalerba P, Cho RW, Clarke MF. Cancer stem cells: models and concepts. Annu Rev Med. 2007;58:267-84. doi: 10.1146/annurev.med.58.062105.204854. PMID 17002552
- [Background] Sanli T, Storozhuk Y, Linher-Melville K, Bristow RG, Laderout K, Viollet B, Wright J, Singh G, Tsakiridis T. Ionizing radiation regulates the expression of AMP-activated protein kinase (AMPK) in epithelial cancer cells: modulation of cellular signals regulating cell cycle and survival. Radiother Oncol. 2012 Mar;102(3):459-65. doi: 10.1016/j.radonc.2011.11.014. Epub 2012 Jan 5. PMID 22225791
- [Background] Eyler CE, Foo WC, LaFiura KM, McLendon RE, Hjelmeland AB, Rich JN. Brain cancer stem cells display preferential sensitivity to Akt inhibition. Stem Cells. 2008 Dec;26(12):3027-36. doi: 10.1634/stemcells.2007-1073. Epub 2008 Sep 18. PMID 18802038
- [Background] Song CW, Lee H, Dings RP, Williams B, Powers J, Santos TD, Choi BH, Park HJ. Metformin kills and radiosensitizes cancer cells and preferentially kills cancer stem cells. Sci Rep. 2012;2:362. doi: 10.1038/srep00362. Epub 2012 Apr 12. PMID 22500211